CLINICAL TRIAL: NCT00468806
Title: An Open Label Positron Emission Tomography Study in Healthy Male Subjects to Investigate Brain Dopamine D3 Occupancy Kinetics, Pharmacokinetics and Safety of Single Oral Doses of GSK598809, Using [11C]-(+)-PHNO as PET Ligand.
Brief Title: Study of Safety, Blood Levels and Brain Receptor Occupancy of GSK598809 Using PET Imaging in Health Males.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DAN106589
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Healthy Subjects
Keywords: PET scan; Health Males
MeSH Terms: interventions — GSK598809; naxagolide

INTERVENTIONS:
Drug: GSK598809, using [11C]-(+)-PHNO

SUMMARY:
The purpose of this study is to look at how much of a new drug, GSK598809 binds to specific proteins in the brain and how much stays in the blood over a range of different doses.

ELIGIBILITY:
Inclusion Criteria:

Healthy male subjects, defined as individuals who are free from clinically significant illness or disease as determined by their medical history (including family), physical examination, laboratory studies, and other tests.

* Aged 25-55 years inclusive, at screening visit.
* Body weight > 50 kg and body mass index (BMI) between 19.0 - 29.0 kg/m2 inclusive.
* Capable of giving informed consent and can comply with the study requirements and timetable.
* Self-administered Beck Depression Inventory II scale total score no greater than 9, and suicide question score of zero.
* Able to read, comprehend and record information.
* A signed and dated written informed consent is obtained from the subject.

Exclusion Criteria:

* The physician responsible considers the subject unfit for the study based upon medical history, physical examination and psychiatric history and evaluation.
* History of a drug or other allergy which in the opinion of the physician responsible contraindicates their participation in the study.
* Participation in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug(whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* A screening ECG outside of ranges specified in the protocol
* Pulse rate <55 or >100 bpm OR a systolic blood pressure >140 and <100 OR a diastolic blood pressure >90 and <60.
* History of long QT syndrome (personal or family) or other cardiac conduction disorder, or other clinically significant cardiac disease.
* An electrolyte value outside the normal range at pre-study screening. Subjects who do not fall within the normal reference ranges may be included within the study if in the opinion of the Principal Investigator and Medical Monitor this will not compromise the subject.
* Liver function tests (LFT) elevated above the reference range at pre-study screening that remain elevated with a repeat LFT.
* Any other clinically significant laboratory abnormality.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John'sWort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption averaging >14 drinks/week for men. One drink is equivalent to(12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits) within 6 months of screening.
* Smokes or has smoked in the last 6 months.
* Donation of more than 450 ml blood within the 56 days before dosing.
* An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women from the time of administration of study medication (GSK598809) until 90 days following administration of study medication or an unwillingness of the male subject to use a condom/spermicide in addition to having their female partner use another form of contraception if the woman could become pregnant from the time of administration of study medication until 90 days following administration of study medication.
* Current or recent (within one year) gastrointestinal disease; a history of malabsorption, esophageal reflux, irritable bowel syndrome; frequent (more than once a week) occurrence of heartburn; or any surgical intervention (e.g., cholecysectomy) which would be expected to influence the absorption of drugs.
* Any previous or current psychiatric diagnosis listed in DSMIV Axis I or II.
* Any history of suicidal attempts, suicidal ideation or behaviour.
* Chronic Hepatitis B and C, as evidenced by positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody.
* A positive test for HIV.
* Past history of drug abuse (i.e. meeting DSM IV or ICD 10 criteria for substance dependence) or has tested positive for urine drugs of abuse at pre-study screening and/or prior to dosing.
* Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden (a significant radiation burden being defined as ICRP category IIb or above: No more than 10 mSv in addition to natural background radiation, in the previous 3 years including the dose from this study).
* Family history of cancer (one or more first-degree relative diagnosed before the age of 55).
* History of or suffers from claustrophobia or feels that they will be unable to lie still on their back in the PET camera for a period of 2 hours.
* History or presence of a neurological diagnosis (not limited to but including for example, stroke, traumatic brain injury, epilepsy, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischemic attack, schizophrenia, major depression etc) that may influence the outcome or analysis of the scan results.
* Presence of a cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies as assessed by a standard pre-MRI.

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
%D3 RO at Tmax | approx 1.5 hrs
Percentage occupancy at Tmax | approx 1.5 hrs
Ttrough | approx 24 hrs
time course of GSK598809 plasma concentration following a single oral dose of GSK598809 | at predose,1,1.5,2,3,4,8,24 and 48 hrs.

SECONDARY OUTCOMES:
Prolactin/TSH levels | at predose,1, 2, 4,8 & 24 hrs postdose
Akathisia | at baseline at 1, 4 hrs postdose
EPQ, BIS-BAS: | at screening
POMS, CRT: | at predose & 4 hrs postdose
VAS: | at predose, 1, 4 hrs postdose
LSEQ | at screening, baseline scan & 24 hrs
neuroendocrine and behavioural measures following GSK598809 administration.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Searle G, Beaver JD, Comley RA, Bani M, Tziortzi A, Slifstein M, Mugnaini M, Griffante C, Wilson AA, Merlo-Pich E, Houle S, Gunn R, Rabiner EA, Laruelle M. Imaging dopamine D3 receptors in the human brain with positron emission tomography, [11C]PHNO, and a selective D3 receptor antagonist. Biol Psychiatry. 2010 Aug 15;68(4):392-9. doi: 10.1016/j.biopsych.2010.04.038. PMID 20599188